CLINICAL TRIAL: NCT02757144
Title: A Dose Block-randomized, Double-blind, Placebo- and Active-controlled, Single and Multiple Dosing, Dose-escalation Clinical Phase 1 Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DWP14012 After Oral Administration in Healthy Male Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DWP14012 After Oral Administration in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DW_DWP14012001
Record Dates: First submitted 2016-03-16; First posted 2016-04-29 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Healthy
MeSH Terms: interventions — fexuprazan; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (14):
- Cohort 1: DWP14012 Amg (Experimental): DWP14012 Amg, tablets, orally, single dose administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Cohort 2: DWP14012 Bmg (Experimental): DWP14012 Bmg, tablets, orally, single dose administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Cohort 3: DWP14012 Cmg (Experimental): DWP14012 Cmg, tablets, orally, single dose administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Cohort 4: DWP14012 Dmg (Experimental): DWP14012 Dmg, tablets, orally, single dose administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Cohort 5: DWP14012 Emg (Experimental): DWP14012 Emg, tablets, orally, single dose administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Cohort 6: DWP14012 Fmg (Experimental): DWP14012 Emg, tablets, orally, single dose administration
  Interventions: Drug: DWP14012; Drug: Placebo
- Cohort 1-6: Placebo (Placebo Comparator): DWP14012 placebo-matching tablets, Active-control placebo-matching tablets, orally, single dose administration
  Interventions: Drug: Placebo
- Cohort 1-6: Esomeprazole (Active Comparator): Nexium® tablets, orally, single dose administration
  Interventions: Drug: Placebo; Drug: Esomeprazole
- Cohort 7: DWP14012 Amg (Experimental): DWP14012 Amg, tablets, orally, repeated dose administration(for 7days)
  Interventions: Drug: DWP14012; Drug: Placebo
- Cohort 8: DWP14012 Bmg (Experimental): DWP14012 Bmg, tablets, orally, repeated dose administration(for 7days)
  Interventions: Drug: DWP14012; Drug: Placebo
- Cohort 9: DWP14012 Cmg (Experimental): DWP14012 Cmg, tablets, orally, repeated dose administration(for 7days)
  Interventions: Drug: DWP14012; Drug: Placebo
- Cohort 7-10: Placebo (Placebo Comparator): DWP14012 placebo-matching tablets, Active-control placebo-matching tablets, orally, repeated dose administration(for 7days)
  Interventions: Drug: Placebo
- Cohort 7-10: Esomeprazole (Active Comparator): Nexium®, orally, repeated dose administration(for 7days)
  Interventions: Drug: Placebo; Drug: Esomeprazole
- Cohort 9: DWP14012 Dmg (Experimental): DWP14012 Dmg, tablets, orally, repeated dose administration(for 7days)
  Interventions: Drug: DWP14012; Drug: Placebo

INTERVENTIONS:
Drug: DWP14012 — DWP14012 tablets
  Arms: Cohort 1: DWP14012 Amg; Cohort 2: DWP14012 Bmg; Cohort 3: DWP14012 Cmg; Cohort 4: DWP14012 Dmg; Cohort 5: DWP14012 Emg; Cohort 6: DWP14012 Fmg; Cohort 7: DWP14012 Amg; Cohort 8: DWP14012 Bmg; Cohort 9: DWP14012 Cmg; Cohort 9: DWP14012 Dmg
Drug: Placebo — DWP14012 placebo-matching tablets, Active control placebo-matching tablets
Drug: Esomeprazole — Nexium®
  Arms: Cohort 1-6: Esomeprazole; Cohort 7-10: Esomeprazole

SUMMARY:
This is a dose block-randomized, double-blind, placebo- and active-controlled, single and multiple dosing, dose-escalation clinical phase 1 trial to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of DWP14012 after oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged between 19 and 50 at screening
* Those whose weight is between 55 and 90 kg and BMI is between 18.0 and 27.0
* Those who are adequate to be subjects in this study upon judgment of the investigator after physical examination, clinical laboratory test, examination by interview, etc

Exclusion Criteria:

* Those who have clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history
* Those who have gastrointestinal diseases or past history of gastrointestinal diseases (gastrointestinal ulcer, gastritis, gastrospasm, gastroesophageal reflux, Crohn's disease etc.) that may affect safety and pharmacokinetic/pharmacodynamic evaluation of study drug, and those who have past history of gastrointestinal surgery (however, except simple appendectomy and herniotomy)
* Those who have been Helicobacter pylori positive
* Those whose plasma AST (SGOT) and ALT (SGPT) exceed 1.5 times to the upper limit of the normal range in screening including additional examinations prior to randomization
* Those who have anatomical disability in insertion and maintenance of pH meter catheter

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number and percentage of Participants With Adverse Events (AE) | Day -2(Randomization) to Day 11~18(Post-study visit)
  All AE standardized using MedDRA was assessed by investigator using the protocol defined grading system. Intensity was categorized as mild, moderate adn severe.
Number and percentage of Participants With Adverse Drug Reactions (ADR) | Day -2(Randomization) to Day 11~18(Post-study visit)
  An adverse drug reaction (ADR) is an injury caused by taking an investigational product.
Number of Participants With Clinically Significant Vital Sign findings | Day -2(Randomization) to Day 11~18(Post-study visit)
  Blood pressure, pulse and body temperature were tested. The Average, Median, Standard Deviation, Min, Max values will be calculated to assess the safety/tolerability.
Number of Participants With Clinically Significant Electrocardiogram(12-lead ECG) findings | Day -2(Randomization) to Day 11~18(Post-study visit)
  Ventricular rate, RR interval, PR interval, QRS duration, QTcB and QTcF were recorded. The results of 12-lead ECG will be categorized Normal/Abnormal NCS(No clinically significant)/Abnormal CS(clinically significant).
Number of Participants With Clinically Significant Laboratory results | Day -2(Randomization) to Day 11~18(Post-study visit)
  Hematology, Blood chemistry, Coagulation and Urinalysis were tested. The Average, Median, Standard Deviation, Min, Max values will be calculated to assess the safety/tolerability.

SECONDARY OUTCOMES:
Cmax: Maximum concentration of DWP14012 | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours
  in single ascending dose cohort
Cmax,ss: Maximum concentration of DWP14012 at steady state | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24h, Day 3-6 pre-dose, Day 7 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours
  in multiple ascending dose cohort
Cmin,ss: Minimum concentration of DWP14012 at steady state | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24h, Day 3-6 pre-dose, Day 7 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours
  in multiple ascending dose cohort
Tmax: Time of maximum concentration | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours
  in single ascending dose cohort
Tmax,ss: Time of maximum concentration at steady state | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24h, Day 3-6 pre-dose, Day 7 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours
  in multiple ascending dose cohort
AUClast: Area under the plasma concentration-time curve from time 0 to 48hours | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours
  in single ascending dose cohort
AUCinf: Area under the plasma concentration-time curve from time 0 to infinity | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours
  in single ascending dose cohort
AUCtau: Area under the plasma concentration-time curve from time 0 to tau(dosing interval) | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24h, Day 3-6 pre-dose, Day 7 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours
  in multiple ascending dose cohort
T1/2: Elimination half-life | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours
  in single ascending dose cohort
T1/2: Elimination half-life | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24h, Day 3-6 pre-dose, Day 7 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours
  in multiple ascending dose cohort
Percentage of total time that the intragastric pH was above 4 | Day 1
  After single administration of the investigational products, 24hr gastric pH monitoring started.
Percentage of total time that the intragastric pH was above 4 | Day 7
  After multiple administration of the investigational products, 24hr gastric pH monitoring started.
Serum gastrin concentration profile | Day -2(Randomization) to Day 11~18(Post-study visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea